CLINICAL TRIAL: NCT07213336
Title: Effect of Trigger Point Massage and Stretching Exercises on Menstruation Symptoms, Pain Intensity and Quality of Life in Primary Dysmenorrhea
Brief Title: A New Treatment for Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Zeynep İrem Kar, specialist physiotherapist, Halic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HalicU-FTR-ZİK-01
Record Dates: First submitted 2025-09-17; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Primary Dysmenorrhea (PD)
Keywords: Stretching exercises; menstrual pain; primary dysmenorrhea; trigger point massage
MeSH Terms: conditions — Dysmenorrhea | interventions — Exercise; Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. group (No Intervention): Control group
- 2.group (Experimental): Stretching exercise group
  Interventions: Other: Exercise, massage
- 3.group (Experimental): trigger point massage and stretching exercise group
  Interventions: Other: Exercise, massage

INTERVENTIONS:
Other: Exercise, massage — trigger point massage and stretching exercise
  Arms: 2.group; 3.group

SUMMARY:
Primary dysmenorrhea (PD) is a chronic health condition that affects primarily young women and interferes with daily activities, causes loss of work productivity, and reduces quality of life. In this controlled study, the effects of trigger point massage and stretching exercises applied to patients diagnosed with primary dysmenorrhea on pain severity (Visual Analog Scale), menstrual symptoms (Menstruation Symptom Scale) and quality of life (SF-36) were investigated. Forty-five women who were followed up with the diagnosis of Primary Dysmenorrhea in the Gynecology and Obstetrics Clinic of a local Hospital. Participants were randomly assigned to exercise, exercise+trigger point, and control groups using a computer-generated randomization list. The "Visual Analog Scale" was used to evaluate the severity of menstrual pain, "Menstruation Symptom Scale" was used to evaluate the severity of menstrual symptoms, and "SF-36" was used to evaluate the quality of life.

DETAILED DESCRIPTION:
This controlled experimental study included 45 volunteers diagnosed with primary dysmenorrhea by a gynecologist. Participants were randomly assigned to three groups using the "Research Randomizer" web program. The control group (n=14) received no intervention. The stretching exercise group (n=15) received only stretching exercises; the stretching and trigger point group (n=15) received stretching exercises plus trigger point massage of the quadratus lumborum, rectus abdominus, iliopsoas, and hip adductor muscles, all performed by the same trained physiotherapist.

Study Inclusion Criteria:

* Being a woman between the ages of 18 and 30,
* Having a diagnosis of primary dysmenorrhea,
* Being a nulliparous,
* Having a regular menstrual cycle (28 ± 7 days). Exclusion Criteria
* Having rheumatic, gastrointestinal, psychiatric, surgical, or other chronic pain syndromes;
* Being on any anti-inflammatory, analgesic, or non-convertible progestin pill (OCP) Participants in the control group were not included in the treatment program administered to the other participants for 8 weeks, but continued the NSAID medication prescribed by the doctor who diagnosed dysmenorrhea.

Participants in the stretching group underwent a 45-minute exercise program twice a week, accompanied by a physiotherapist, for 8 weeks. Participants in the stretching exercises and trigger point massage group underwent a 45-minute exercise program twice a week, accompanied by a physiotherapist, for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 18 and 30
* Having a diagnosis of primary dysmenorrhea
* Not having given birth
* Having a regular menstrual cycle (28 ± 7 days)

Exclusion Criteria:

* Having been diagnosed with rheumatic, gastrointestinal, psychiatric, neurological diseases, or other chronic pain syndromes
* Being on any anti-inflammatory, analgesic, or estrogen/progestin pill (OCP) treatment

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 44 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
SF-36 | The 1st and 3rd Most Painful Days of the Menstrual Cycle
  SF-36: This questionnaire has 8 subscales, totaling 36 questions: 10 items on "physical function," 7 items on "role limitations due to physical (4 items) and emotional problems (3 items), 2 items on "pain," 4 items on "vitality," 2 items on "social function," 5 items on "mental health," and 5 items on "general health.
Visual Analog Scale | The 1st and 3rd Most Painful Days of the Menstrual Cycle
  Visual Analog Scale: The visual analog scale (VAS) is the most commonly used tool for assessing pain intensity. It is easy to use, provides reproducible results, and can be applied to a variety of practice settings.
Personal Information Form | The 1st and 3rd Most Painful Days of the Menstrual Cycle
  Personal Information Form: This form includes personal information.
menstrual symptom scale | The 1st and 3rd Most Painful Days of the Menstrual Cycle
  It consists of a 5-point Likert-type scale with a total of 24 items. Individuals are asked to rate their menstruation-related symptoms between 1 (never) and 5 (always). The MBI score is calculated by averaging the total scores of the scale items. A higher mean score indicates an increased severity of menstrual symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: melek g yavuzer, Study Director
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want it to be shared without being published in any journal.

DOCUMENTS (1):
  • Informed Consent Form (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT07213336/ICF_000.pdf